CLINICAL TRIAL: NCT00230932
Title: Validation of Pain as a Vital Sign Among Veterans With Advanced Illness
Brief Title: Help Veterans Experience Less Pain Study (HELP-Vets)
Acronym: HELP-Vets
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 03-150
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-11

CONDITIONS: Pain; Heart Failure, Congestive; Signs and Symptoms
Keywords: Veterans; Pain; Palliative Care; Cardiology; Reproducibility of Results; Health Personnel; Heart Failure, Congestive
MeSH Terms: conditions — Pain; Heart Failure; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: outpatients selected from random visits in primary care, oncology, and cardiology clinics

SUMMARY:
Our purpose is to evaluate the reliability and validity of the '5th vital sign' in everyday practice settings and to compare the relationship of pain to other symptoms and pain treatment in patients with cancer, CHF, and patients with complex general medical illness and poor self-reported health.

DETAILED DESCRIPTION:
Background/Rationale: The Veterans Administration (VA) faces a substantial challenge in trying to improve symptomatic care. An important priority is how to ensure pain relief. Studies show that pain is a major symptom for patients with advanced chronic illness in general. Drawing upon different clinical paradigms for the evaluation and treatment of pain, this study focuses on improving measurement and interpretation of routine pain screening in ambulatory VA patients as an important step to improving end-of-life care. Objective(s): In a variety of outpatient settings (hospital-based, large outpatient multi-specialty, and community-based) at the VA Greater Los Angeles (GLA) and Long Beach (LB) Healthcare Systems, we conducted surveys to capture patient, nurse, and clinician perspectives to evaluate the reliability and validity of pain as a 5th vital sign. We assessed skills that may be associated with pain measurement practices of nursing staff. Clinician knowledge, attitudes, and behaviors regarding the need to alleviate pain detected on routine screening were evaluated. Methods: Screen, enroll, and survey 650 cognitively intact patients with advanced CHF, cancer, and advanced general medical illness stratified by self-reported health status immediately after they are seen in outpatient clinics (general medicine, oncology, and cardiology clinics). Patients were approached and surveyed immediately after the outpatient visit on validated pain instruments, measures of depression, other symptoms, quality of life, attitudinal barriers to treatment of pain, the pain rating process, and unmet needs and satisfaction with treatment of pain, depression, and other symptoms. All nursing staff working as pain raters in the general medicine, oncology, and cardiology clinics were surveyed to assess relevant skills that may be associated with pain measurement practices. All clinicians (physicians, nurse practitioners, and physician assistants) working as treatment providers in these clinics were surveyed after patient visits to assess knowledge, attitudes, and behaviors of clinicians with regard to the need to alleviate pain detected on routine screening. Results: We found that in approximately 50% of cases, clinic staff taking vital signs used informal (e.g., 'How do you feel?') rather than forma (e.g., 0-10 NRS) methods to assess pain, and that practice was associated with underestimation of patient-reported pain to research staff in about 30% of cases. Factors associated with underestimation of patient reported pain to nurses compared with research raters included more years of staff work experience, patient anxiety or PTSD disorders, and lower self-reported health. Overestimation was associated with adherence to the formal NRS and negatively associated with a better environment for pain rating. About 40% of patients had emotional distress which was higher among patients in moderate to severe pain (62%). Only prior diagnosis and sleep interference due to pain were associated with provider detection of distress. Status: Enrollment is closed; IRB approved at VA GLA and LB Healthcare Systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking care in VA outpatient primary care, oncology, cardiology, or community based outpatient clinics, for advanced cancer, congestive heart failure, and advanced, complex general medical illness stratified by self-reported health.
* Patients will be screened for fair or poor general medical health status, health conditions (cancer, CHF), cognition and ability to complete a researcher-assistant guided survey (e.g., hearing intact).
* All nursing staff and pain treatment staff (resident and staff physician, PA, NP) in general medicine, oncology, and cardiology care at selected study sites and related community-based clinics will be asked to participate.

Exclusion Criteria:

* Patients who are hearing and/or cognitively impaired.
* Patients who do not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 654 veterans, 50% with fair to poor, and 50% with good to excellent self-reported health
Sampling Method: Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2005-10; Primary Completion 2007-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
patient reported pain to nurses (NRS) compared to research raters (NRS, BPI) | cross sectional, visit based

CONTACTS AND LOCATIONS:
Overall Officials: Karl A. Lorenz, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Lorenz KA, Shugarman LR, Lynn J. Health care policy issues in end-of-life care. J Palliat Med. 2006 Jun;9(3):731-48. doi: 10.1089/jpm.2006.9.731. No abstract available. PMID 16752979
- [Result] Walling AM, Asch SM, Lorenz KA, Roth CP, Barry T, Kahn KL, Wenger NS. The quality of care provided to hospitalized patients at the end of life. Arch Intern Med. 2010 Jun 28;170(12):1057-63. doi: 10.1001/archinternmed.2010.175. PMID 20585072
- [Result] Shugarman LR, Asch SM, Meredith LS, Sherbourne CD, Hagenmeier E, Wen L, Cohen A, Rubenstein LV, Goebel J, Lanto A, Lorenz KA. Factors associated with clinician intention to address diverse aspects of pain in seriously ill outpatients. Pain Med. 2010 Sep;11(9):1365-72. doi: 10.1111/j.1526-4637.2010.00931.x. Epub 2010 Aug 30. PMID 20807347
- [Result] Goebel JR, Sherbourne CD, Asch SM, Meredith L, Cohen AB, Hagenmaier E, Lanto AB, Simon B, Rubenstein LV, Shugarman LR, Lorenz KA. Addressing patients' concerns about pain management and addiction risks. Pain Manag Nurs. 2010 Jun;11(2):92-8. doi: 10.1016/j.pmn.2009.03.009. Epub 2009 Sep 12. PMID 20510839
- [Result] Shugarman LR, Goebel JR, Lanto A, Asch SM, Sherbourne CD, Lee ML, Rubenstein LV, Wen L, Meredith L, Lorenz KA. Nursing staff, patient, and environmental factors associated with accurate pain assessment. J Pain Symptom Manage. 2010 Nov;40(5):723-33. doi: 10.1016/j.jpainsymman.2010.02.024. Epub 2010 Aug 8. PMID 20692807
- [Result] Stone SC, Mohanty SA, Gruzden C, Lorenz KA, Asch SM. Emergency department research in palliative care: challenges in recruitment. J Palliat Med. 2009 Oct;12(10):867-8. doi: 10.1089/jpm.2009.0139. No abstract available. PMID 19807230
- [Result] Grudzen CR, Koenig WJ, Hoffman JR, Boscardin WJ, Lorenz KA, Asch SM. Potential impact of a verbal prehospital DNR policy. Prehosp Emerg Care. 2009 Apr-Jun;13(2):169-72. doi: 10.1080/10903120802471923. PMID 19291552
- [Result] Seow H, Snyder CF, Mularski RA, Shugarman LR, Kutner JS, Lorenz KA, Wu AW, Dy SM. A framework for assessing quality indicators for cancer care at the end of life. J Pain Symptom Manage. 2009 Dec;38(6):903-12. doi: 10.1016/j.jpainsymman.2009.04.024. PMID 19775860
- [Result] Grudzen CR, Timmermans S, Koenig WJ, Torres JM, Hoffman JR, Lorenz KA, Asch SM. Paramedic and emergency medical technicians views on opportunities and challenges when forgoing and halting resuscitation in the field. Acad Emerg Med. 2009 Jun;16(6):532-8. doi: 10.1111/j.1553-2712.2009.00427.x. Epub 2009 May 11. PMID 19438412
- [Result] Goebel JR, Doering LV, Shugarman LR, Asch SM, Sherbourne CD, Lanto AB, Evangelista LS, Nyamathi AM, Maliski SL, Lorenz KA. Heart failure: the hidden problem of pain. J Pain Symptom Manage. 2009 Nov;38(5):698-707. doi: 10.1016/j.jpainsymman.2009.04.022. Epub 2009 Sep 3. PMID 19733032
- [Result] Zubkoff L, Lorenz KA, Lanto AB, Sherbourne CD, Goebel JR, Glassman PA, Shugarman LR, Meredith LS, Asch SM. Does screening for pain correspond to high quality care for veterans? J Gen Intern Med. 2010 Sep;25(9):900-5. doi: 10.1007/s11606-010-1301-5. Epub 2010 Mar 14. PMID 20229139
- [Result] Lorenz KA, Krebs EE, Bentley TG, Sherbourne CD, Goebel JR, Zubkoff L, Lanto AB, Asch SM. Exploring alternative approaches to routine outpatient pain screening. Pain Med. 2009 Oct;10(7):1291-9. doi: 10.1111/j.1526-4637.2009.00709.x. PMID 19818039
- [Result] Sherbourne CD, Asch SM, Shugarman LR, Goebel JR, Lanto AB, Rubenstein LV, Wen L, Zubkoff L, Lorenz KA. Early identification of co-occurring pain, depression and anxiety. J Gen Intern Med. 2009 May;24(5):620-5. doi: 10.1007/s11606-009-0956-2. Epub 2009 Mar 24. PMID 19308333
- [Result] Goebel JR, Doering LV, Evangelista LS, Nyamathi AM, Maliski SL, Asch SM, Sherbourne CD, Shugarman LR, Lanto AB, Cohen A, Lorenz KA. A comparative study of pain in heart failure and non-heart failure veterans. J Card Fail. 2009 Feb;15(1):24-30. doi: 10.1016/j.cardfail.2008.09.002. Epub 2008 Nov 13. PMID 19181290
- [Result] Cadogan MP, Edelen MO, Lorenz KA, Jones M, Yosef J, Hascall T, Simon B, Harker JO, Ferrell B, Saliba D. The relationship of reported pain severity to perceived effect on function of nursing home residents. J Gerontol A Biol Sci Med Sci. 2008 Sep;63(9):969-73. doi: 10.1093/gerona/63.9.969. PMID 18840802
- [Result] Lorenz KA, Sherbourne CD, Shugarman LR, Rubenstein LV, Wen L, Cohen A, Goebel JR, Hagenmeier E, Simon B, Lanto A, Asch SM. How reliable is pain as the fifth vital sign? J Am Board Fam Med. 2009 May-Jun;22(3):291-8. doi: 10.3122/jabfm.2009.03.080162. PMID 19429735
- [Result] Dy SM, Asch SM, Lorenz KA, Weeks K, Sharma RK, Wolff AC, Malin JL. Quality of end-of-life care for patients with advanced cancer in an academic medical center. J Palliat Med. 2011 Apr;14(4):451-7. doi: 10.1089/jpm.2010.0434. Epub 2011 Mar 10. PMID 21391819
- [Result] Riopelle D, Wagner GJ, Steckart J, Lorenz KA, Rosenfeld KE. Evaluating a palliative care intervention for veterans: challenges and lessons learned in a longitudinal study of patients with serious illness. J Pain Symptom Manage. 2011 Jun;41(6):1003-14. doi: 10.1016/j.jpainsymman.2010.09.023. Epub 2011 Mar 12. PMID 21402457
- [Result] Malin JL, O'Neill SM, Asch SM, Dy SM, Walling AM, Tisnado D, Antonio AL, Lorenz KA. Quality of supportive care for patients with advanced cancer in a VA medical center. J Palliat Med. 2011 May;14(5):573-7. doi: 10.1089/jpm.2010.0464. Epub 2011 Mar 17. PMID 21413885